CLINICAL TRIAL: NCT03656757
Title: The Impact of Altered Arterioventricular Coupling on Central Cardiovascular Energy Delivery
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/767
Record Dates: First submitted 2018-08-31; First posted 2018-09-04 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiac Power; Oscillatory Power; Coronary Artery Bypass Graft; Arterioventricular Coupling
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will assess the amount of energy that the heart will deliver to the central circulation and the efficiency of that energy transfer, in patients undergoing a coronary artery bypass graft operation. Measurements will be taken just after induction of anaesthesia and repeated just after the end of the operation. The total energy delivered by the heart will be calculated by multiplying a pressure curve from the artery in the hand with the instantaneous ultrasound recorded cardiac output flow curve. The energy responsible for the acceleration of the blood volume, known as oscillatory power will also be calculated. The energy transfer will be calculated using a mathematical model based upon other ultrasound and blood pressure recorded variables. We would like to see if any alteration in energy delivered is in part due to impairment in energy transfer or alteration of fraction of oscillatory power rather than a change in total energy production. We would also like to study if there are changes in the oscillatory power after cardiac bypass surgery. The patients will be sampled sequentially into the study. We are not aware of any such studies undertaken in humans previously.

ELIGIBILITY:
Inclusion Criteria:

* Elective Coronary Artery Bypass Graft patients
* No contraindications to transoesophageal Echo
* Ejection fraction 40% or over

Exclusion Criteria:

* Lack of consent
* Emergency operation
* Prosthetic aortic valve

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population undergoing elective coronary artery bypass grafting typically have multiple cardiovascular risk factors such as hypertension, hyperlipidaemia, diabetes and smoking.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-03-13 (Actual); Study Completion 2019-03-13 (Actual)

PRIMARY OUTCOMES:
Arterioventricular coupling | 1 day
  The ratio between arterial elastance and ventricular elastance
Total Cardiac Power | 1 day
  The amount of energy per second delivered from the left ventricle to the arterial circulation
Oscillatory Cardiac Power | 1 day
  The part of total cardiac power which is responsible for acceleration of the blood volume during systole.

SECONDARY OUTCOMES:
Cardiac Output | 1 day
  The hearts delivery of volume per minute
Heart rate | 1 day
  The amount of heart beats per minute
Systemic vascular resistance | 1 day
  The resistance to flow of the arterial tree

CONTACTS AND LOCATIONS:
Overall Officials: Idar Kirkeby-Garstad, md phd, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- St Olavs Hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: No